CLINICAL TRIAL: NCT07090863
Title: Additively (AM) Versus Subtractively (SM) Manufactured Implant Supported Fixed Dental Prostheses (iFDPs)
Brief Title: Additively Versus Subtractively Manufactured Implant Supported Fixed Dental Prostheses
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard Medical School (HMS and HSDM) (Other)
Collaborators: University of Zurich (Other)
Responsible Party: Principal Investigator, German O. Gallucci, Professor, Harvard Medical School (HMS and HSDM)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3DP-Implant-Crown
Record Dates: First submitted 2025-07-08; First posted 2025-07-29 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Dental Prosthesis, Implant-Supported
Keywords: 3D-printing; implant-supported prostheses; additive manufacturing

STUDY DESIGN:
Intervention Model Description: Randomised controlled clinical trial
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Additive manufacturing (Experimental): additively manufactured implant-supported prostheses
  Interventions: Device: AM manufacturing method
- Subtractive manufacturing (Active Comparator): subtractively manufactured implant-supported prostheses
  Interventions: Device: SM manufacturing method

INTERVENTIONS:
Device: AM manufacturing method — additively manufactured implant-supported prostheses
  Arms: Additive manufacturing
Device: SM manufacturing method — subtractively manufactured implant-supported prostheses
  Arms: Subtractive manufacturing

SUMMARY:
This research is being done to evaluate the clinical, technical, biological, and aesthetic results of two different fabrication methods (additive and subtractive) for creating implant-supported fixed dental prostheses (iFDPs). Patients will receive an iFDP, meaning an implant-supported crown, according to regular treatment protocols. The fabrication method used to create the implant-supported crown will be decided in a randomised way. Clinical and radiological examinations will be performed prior to and when receiving the implant-supported crown and during a follow-up period of 3 years. Furthermore, technician- and patient-reported outcomes will be evaluated used questionnaires.

DETAILED DESCRIPTION:
This study is designed as a randomised controlled clinical trial with a multi-centre design. Patients in need of a definitive posterior implant-supported crown will be enrolled in this study following predefined eligibility criteria at two different study centres (Harvard School of Dental Medicine, Harvard University and Center of Dental Medicine, University of Zurich). Patients will receive a single implant-supported crown fabricated according to group allocation (additively or subtractively manufactured). After crown delivery, patients will be followed-up for an observation period of 3 years. The primary outcome is the clinical performance of the implant crowns. Clinical, technical, biological, and aesthetic results as well as the technician- and patient-reported outcomes will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form in English language
* ≥ 20 years of age
* In need of at least one definitive screw retained premolar or molar iFDP on an existing dental implant (Straumann AG)
* Presence of at least one adjacent tooth at the implant site
* Adequate oral hygiene
* Capability to comply with the study procedures

Exclusion Criteria:

* Pregnant or lactating women
* Known or suspected non-compliance, drug or alcohol abuse
* Severe periodontal and peri-implant disease

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-07-30 (Estimated); Primary Completion 2029-07-20 (Estimated); Study Completion 2029-07-20 (Estimated)

PRIMARY OUTCOMES:
Clinical success | This outcome will be evaluated at the baseline and at the follow-up visits after 1 year, 2 years and 3 years
  The primary outcome is clinical success of the iFDPs, which is defined as the iFDPs being free of all complications over the entire observation period.

SECONDARY OUTCOMES:
Efficiency during manufacturing (dental technician) (time) | Periprocedural
  Fabrication time for the iFDP will be measured in minutes. The time needed for the manufacturing (subtractively or additively), the post-processing and the cementation on to the titanium base will be measured using a stopwatch.
Efficiency during manufacturing | Periprocedural
  The laboratory workflow during manufacturing will be assessed by the dental technicians using a questionnaire on success of the fabrication and postprocessing steps, and complications such as faulty/damaged iFDP. Dental technicians will report complications by answering yes/no to the occurrence of any complications, specifying occurred complications and reporting their quantity.
Chairside adjustment time | Periprocedural
  The total mean time for chairside adjustment (min) at iFDP delivery. A stopwatch will be used to measure the minutes between removing the healing abutment of the implant and final insertion of the prostheses after finishing any potential adjustments (for example approximal/occlusal contacts, polishing)
Survival rate | This outcome will be reported on the baseline visit and the follow-up visits after 1, 2 and 3 years
  Survival will be defined as the presence of the iFDP independent of technical, biological or aesthetic complications.
Probing Depth | This outcome will be assessed at the baseline visit and the follow-up visits after 1, 2 and 3 years.
  Measured from the gingival margin to the bottom of the probable pocket to the nearest millimeter using a University of North Carolina (UNC15) periodontal probe with 1 mm markings (Hu-Friedy, Chicago, IL. USA) with a light probing force (≃ 0.2 N)
Esthetic outcomes | This outcome will be assessed at the baseline visit and the follow-up visits after 1, 2 and 3 years.
  Standardized photographs, occlusal and buccal aspect will be taken from each patient at each visit for documentation purposes and for evaluating the esthetic aspects. Outcomes will be assessed by using modified criteria of United States Public Health Services (USPHS) (Barnes, Arpante et al. 1995).
Technical outcomes | this outcome will be assessed at the baseline visit and the follow-up visits after 1, 2 and 3 years.
  Technical outcomes of the iFDP will be assessed using modified criteria of United States Public Health Services (USPHS) (Barnes, Arpante et al. 1995).
Patient-reported outcomes | This outcome will be assessed at the baseline and follow-up visits after 1, 2 and 3 years
  Patient satisfaction to the treatment and iFDP will be assessed with questions on Visual Analogue Scale (VAS). Patients will be asked questions regarding their satisfaction on a scale of 0 (not satisfied) to 100 (very satisfied) with the prostheses.
Adverse events | through study completion. This outcome will be reported at baseline and follow-up visits after 1, 2 and 3 years.
  Any Adverse Event (AE) related or possibly related to the study procedures.
Bleeding on probing (BOP) | This outcome will be assessed at the baseline visit and the follow-up visits after 1, 2 and 3 years.
  Presence of bleeding within 30 s after gently probing. The percentage of positive answers will be calculated.
Plaque control record | This outcome will be assessed at the baseline visit and the follow-up visits after 1, 2 and 3 years.
  Presence of plaque evaluated dichotomously. The percentage of positive answers will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: German O Gallucci, Professor, Principal Investigator — Harvard School of Dental Medicine
Locations (2):
- Harvard School of Dental Medicine, Boston, Massachusetts, United States
- Center of Dental Medicine, University of Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
IPD used in the results publication